CLINICAL TRIAL: NCT04471103
Title: Multi-round Compared to Real-Time Delphi for Consensus in Core Outcome Set (COS) Development: A Randomised Trial
Brief Title: Comparison of Multi-Round and Real-Time Delphi Survey Methods
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University of Ireland, Galway, Ireland (Other)
Collaborators: Health Research Board, Ireland (Other)
Responsible Party: Principal Investigator, Prof. Declan Devane, Scientific Director, Health Research Board - Trials Methodology Research Network
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: NUIreland-COHESION
Record Dates: First submitted 2020-07-02; First posted 2020-07-15 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-09

CONDITIONS: Consensus Development
Keywords: Delphi; Real-Time Delphi; Multi-Round Delphi; Randomised Trial; Two-Group Parallel; Survey

STUDY DESIGN:
Intervention Model Description: A two-group parallel randomised trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real-Time Delphi Method (Experimental): The Real-Time Delphi Method involves a single-round Delphi survey rating the importance of outcomes for neonatal encephalopathy. Feedback on each outcome (participant's own rating score, rating of the outcome by stakeholder group and overall consensus results for that outcome) will be provided to the participant once they have rated an outcome. They can then modify how they rated the outcome based on this feedback if they wish. Participants can also re-visit and re-rate outcomes as many times as they wish when the survey is live. Duration will span approximately 5 weeks.
  Interventions: Other: Participation in a Delphi survey
- Multi-round Delphi Method (Active Comparator): The Multi-Round Delphi Method involves a three-round Delphi survey rating the importance of outcomes for neonatal encephalopathy. Feedback on each outcome (participant's own rating score, rating of the outcome by stakeholder group and overall consensus results for that outcome) will be provided to the participant at the end of Round 1 and the end of Round 2. Participants can then modify how they rated the outcome based on feedback, in Rounds 2 and 3, if they wish. Each survey Round will run for 3 weeks approximately. In between survey Rounds, there will be a downtime of approximately 10 days before providing feedback and a further 7 days before starting the next round. Duration will span approximately 14 weeks.
  Interventions: Other: Participation in a Delphi survey

INTERVENTIONS:
Other: Participation in a Delphi survey — Participants will be asked to participate in an online Delphi survey (using one of two randomly allocated methods) to rate the importance of outcomes that should be measured to determine the effect of treatment for neonatal encephalopathy. Outcomes will be prioritised on their importance in a consensus-driven manner.

SUMMARY:
A two-group parallel randomised trial of Delphi survey methods.

DETAILED DESCRIPTION:
Aim:

The aim of this trial is to compare a multi-round Delphi survey method with a Real-Time Delphi method on prioritised outcomes included in a core outcome set (COS). This trial is embedded within the COHESION study which is developing a COS for interventions for the treatment of neonatal encephalopathy.

Methods:

Stakeholders (parents/ caregivers of infants diagnosed and treated with neonatal encephalopathy, healthcare providers and researchers) will be randomised using stratified randomisation to take part in either a multi-round or Real-Time Delphi. Stakeholders will rate the importance of the same set of outcomes in both arms. We will compare the prioritised outcomes at the end of both surveys as well as other parameters such as feedback, initial condition and iteration effects.

ELIGIBILITY:
Inclusion Criteria:

* parents or caregivers of infants that have been diagnosed with and received treatment for neonatal encephalopathy
* healthcare providers including:

  * neonatal nurse practitioners
  * midwives
  * obstetricians
  * neonatologists/paediatricians
  * neonatal/paediatric neurologists
  * general practitioners who provide long-term care for children with neonatal encephalopathy
  * policymakers
* researchers/ academics with expertise in neonatal encephalopathy treatment.

Exclusion Criteria:

• participants not meeting the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2021-08-13 (Actual); Primary Completion 2022-02-07 (Estimated); Study Completion 2022-02-07 (Estimated)

PRIMARY OUTCOMES:
Comparison of outcomes prioritised within each survey arm | End of both surveys (i.e. when the Multi-Round Delphi round 3 has finished and when the Real-Time Delphi has finished at the end of week 5).
  Comparison of outcomes prioritised by respondents at the end of (i) the Real-time and (ii) multi-round Delphi processes. An outcome is judged 'prioritised' based on the proportion of respondents rating the outcome a 7-9 (inclusive) on a 9-point Likert scale (higher scores = higher importance for inclusion in the COS)

SECONDARY OUTCOMES:
Feedback Effect | Through study completion, an average of 14 weeks.
  The feedback effect will tell if the feedback provided to participants resulted in them amending the rating they have to each outcome on the 9-point scale (higher scores= higher importance for inclusion in the COS)
Initial Condition Effect | During the Real-Time Delphi intervention (5 weeks).
  The initial condition effect will capture if early participant's rating for each outcome on the 9-point scale ( higher scores= higher importance for inclusion in the COS) differs to rating given by later participants.
Iteration Effect | Through study completion, an average of 14 weeks.
  The iteration effect will determine if there is a difference in how consensus is achieved on prioritising each outcome or not, between the Multi-Round and the Real-Time Delphi survey arms
Comparison of outcomes prioritised within each survey arm with the final Core Outcome Set | Through study completion, an average of 1 year.
  Comparison of the of outcome headings prioritised at the end of both the Real-Time and Multi-Round Delphi processes with the outcome headings in the final Core Outcome Set.

OTHER OUTCOMES:
Attrition rates | Attrition rates will be recorded at the end of round 1 (week 3) and round 2 (week 9) in the Multi-Round Delphi and at weeks 2 and 4 in the Real-Time Delphi arm.
  Comparison of attrition rates between multi-round and Real-Time Delphi arms.
Frequency of re-visiting the Real-Time Delphi arm | This will be measured when a participant visits the Real-Time Delphi survey and rates the outcomes fully for a second time (between the start of week 1 and the end of week 5).
  Monitoring how often the Real-Time Delphi was re-visited by participants
Usefulness, Satisfaction and Ease of Use of each survey arm | End of both surveys (i.e. when the Multi-Round Delphi round 3 (week 14) has finished and when the Real-Time Delphi has finished at the end of week 5)
  Participants will be asked in a short questionnaire how they found answering each survey using a modified Usefulness, Satisfaction and Ease of use questionnaire on a 7-point Likert Scale where 1= Strongly Disagree and 7=Strongly Agree.

CONTACTS AND LOCATIONS:
Overall Officials: Declan Devane, PhD, Principal Investigator — Health Research Board - Trials Methodology Research Network
Locations (1):
- HRB-TMRN, Galway, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Quirke FA, Battin MR, Bernard C, Biesty L, Bloomfield FH, Daly M, Finucane E, Haas DM, Healy P, Hurley T, Koskei S, Meher S, Molloy EJ, Niaz M, Bhraonain EN, Okaronon CO, Tabassum F, Walker K, Webbe JRH, Parkes MJ, Kirkham JJ, Devane D. Multi-Round versus Real-Time Delphi survey approach for achieving consensus in the COHESION core outcome set: a randomised trial. Trials. 2023 Jul 19;24(1):461. doi: 10.1186/s13063-023-07388-9. PMID 37468987
- [Derived] Quirke FA, Healy P, Bhraonain EN, Daly M, Biesty L, Hurley T, Walker K, Meher S, Haas DM, Bloomfield FH, Kirkham JJ, Molloy EJ, Devane D. Multi-Round compared to Real-Time Delphi for consensus in core outcome set (COS) development: a randomised trial. Trials. 2021 Feb 15;22(1):142. doi: 10.1186/s13063-021-05074-2. PMID 33588938